CLINICAL TRIAL: NCT04054804
Title: Digital Foot Check by Using the D-Foot, a New Software
Acronym: D-Foot2019
Status: Completed | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Ulla Hellstrand Tang, Principal Investigator, Sahlgrenska University Hospital
Other Study IDs: D-Foot 2019
Record Dates: First submitted 2019-07-25; First posted 2019-08-13 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Diabetic Foot; Diabetic Foot Ulcer; Diabetic Foot Ulcer Neuropathic; Neuropathy;Peripheral; Foot Deformities; Foot Callus
Keywords: risk factor; software; orthotics
MeSH Terms: conditions — Diabetic Foot; Neuritis; Foot Deformities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: D-Foot — A digital foot check i assessed by using the software D-Foot.

SUMMARY:
Patients with diabetes should be thoroughly examined before they are provided with insoles and shoes. In the study the feet are examined with the help of a new software, the D-Foot. D-Foot includes questions and surveys.

The aim of the of the study is evaluate how the patients experience the visit at the department of Prosthetics & Orthotics based on the digital foot check.

DETAILED DESCRIPTION:
Patients with diabetes should be thoroughly examined before they are provided with insoles and shoes. The purpose of the foot examination is to determine whether the patient is at risk of developing diabetic foot ulcers (DFU). Risk factors are: neuropathy, peripheral angiopathy, foot deformities, skin pathologies, earlier history of DFU/amputation. With effective control and examination of the feet, foot complications, such as DFU, can be prevented. In the study the feet are examined with the help of a new software, the D-Foot. D-Foot includes questions and surveys.

The aim of the of the study is evaluate how the patients experience the visit at the department of Prosthetics & Orthotics based on the digital foot check.

ELIGIBILITY:
Inclusion Criteria for patients:

* To be diagnosed diabetes
* Age ≥ 18 years
* To understand the Swedish language.

Inclusion Criteria for certified prosthetist & orthotists

* To work at the department
* To be assigned to work with patients with diabetes at risk of developing foot ulcers.
* Have completed the introduction course D-foot

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients being referred to the Department of Prosthetics & Orthotics at Sahlgrenska Univeristy Hospital with the aim to be provided with insoles, shoes to prevent DFU.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
The questionnaire Orthotic and Prosthetic Users Survey (OPUS) will be used. | 2019-2020
  Participants satisfaction with devices and services at the Department of Prosthetics and Orthotics will be evaluated.

SECONDARY OUTCOMES:
Presence of neuropathy (number) | 2019-2020
  From the software, D-Foot, the number of participants having neuropathy will be reported.
Presence of neuropathy (percentage) | 2019-2020
  From the software, D-Foot, the percentage of participants having neuropathy will be reported
Presence of peripheral angiopathy (number ) | 2019-2020
  From the software, D-Foot, the number of participants having peripheral angiopathy will be reported.
Presence of peripheral angiopathy (percentage ) | 2019-2020
  From the software, D-Foot, the percentage of participants having peripheral angiopathy will be reported.
Presence of calluses (number) | 2019-2020
  From the software, D-Foot, the number of participants having calluses will be reported.
Presence of calluses (percentage) | 2019-2020
  From the software, D-Foot, the percentage of participants having calluses will be reported,
Presence of foot deformities (number) | 2019-2020
  From the software, D-Foot, the number of participants having foot deformities eg. hammertoes, hallux valgus will be reported.
Presence of foot deformities (percentage) | 2019-2020
  From the software, D-Foot, the percentage of participants having foot deformities eg. hammertoes, hallux valgus will be reported.
Presence of foot ulcers (number) | 2019-2020
  From the software, D-Foot, the number of participants having foot ulcers will be reported.
Presence of foot ulcers (percentage) | 2019-2020
  From the software, D-Foot, the percentage of participants having foot ulcers will be reported.
Presence of previous foot ulcers (number) | 2019-2020
  From the software, D-Foot, the number of participants with previous foot ulcers will be reported.
Presence of previous foot ulcers (percentage) | 2019-2020
  From the software, D-Foot, the percentage of participants with previous foot ulcers will be reported.
Presence of previous amputation in the lower extremities (number) | 2019-2020
  From the software, D-Foot, the number of participants with previous amputation in the lower extremities will be reported.
Presence of previous amputation in the lower extremities (percentage) | 2019-2020
  From the software, D-Foot, the percentage of participants with previous amputation in the lower extremities will be reported.
System Usability Scale (SUS). The score range from 0-100 and a SUS score above a 68 would be considered above average and anything below 68 is below average. | 2019-2020
  The SUS provides a reliable tool for measuring the usability. It consists of a 10 item questionnaire with five response options for respondents; from Strongly agree to Strongly disagree. SUS allows you to evaluate a wide variety of products and services, including hardware, software, mobile devices, websites and applications. In this setting the aim is to evaluate how certified prosthetists & orthotists experience the use the web program D-Foot when they examine the patients feet?

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Prostetics & Orthotics, Gothenburg, Region Västragötaland, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zugner R, Jarl G, Sundberg L, Tang UH. Experiences of using a digital tool, the D-foot, in the screening of risk factors for diabetic foot ulcers. J Foot Ankle Res. 2022 Dec 13;15(1):90. doi: 10.1186/s13047-022-00594-9. PMID 36514099